CLINICAL TRIAL: NCT00606073
Title: The Influence of Different Concentrations of Glucose in Culture Media(i.e: ISM1 vs. IVF) on Fertilization and Embryo Quality
Brief Title: The Influence of Different Concentrations of Glucose in Culture Media on Fertilization and Embryo Quality
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Dr. Medeia Michaeli, Hillel Yaffe Medical Center
Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HYMC IRB#31/2007
Record Dates: First submitted 2008-01-21; First posted 2008-02-01 (Estimated); Last update posted 2008-02-01 (Estimated); Status verified 2008-01

CONDITIONS: Fertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- I (Active Comparator): IVF Procedure-IVF Medium
  Interventions: Other: Universal IVF Medium + ISM1 Medium
- II (Active Comparator): IVF Procedure - ISM1 Medium
  Interventions: Other: Universal IVF Medium + ISM1 Medium
- III (Active Comparator): ICSI Procedure - IVF Medium
  Interventions: Other: Universal IVF Medium + ISM1 Medium
- IV (Active Comparator): ICSI Procedure - ISM1 Medium
  Interventions: Other: Universal IVF Medium + ISM1 Medium

INTERVENTIONS:
Other: Universal IVF Medium + ISM1 Medium — Sibling oocytes will be equally divided and incubated separately in different 4-well culture dishes containing either IVF medium or ISM1 Medium and while ICSI will be returned to the same culture dish following injection. Fertilization assessment will be performed approximately after 15-20 hours for standard IVF and 12-18 hours post ICSI performance. After assessment, fertilized oocytes from different culture media will be transferred separately into fresh culture dishes containing ISM1 medium only. The zygotes will be incubated until embryo transfer on day 2 or 3. Embryo quality will be assessed according to the morphology of blastomeres as well as it's developmental stage.

SUMMARY:
The aim of this study is to examine whether incubation of human oocytes until pronuclear stage, in different culture media containing high and low concentrations of glucose affect fertilization differently, not only in standard IVF cycles, but also after intracytoplasmatic sperm injection.In addition, we wish to determine whether exposure of oocytes to different concentrations of glucose until pronuclear stage has further effect on embryo quality and development until the blastocyst stage.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing IVF treatment in our clinic during study period

Exclusion Criteria:

* Females older than 40 years
* Patients with less than 6 retrieved oocytes
* Male patients older than 50 years old
* Patients after testis biopsies

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2008-02; Primary Completion 2009-08 (Estimated)

PRIMARY OUTCOMES:
Fertilization rate and embryo quality | 6 days